CLINICAL TRIAL: NCT00196365
Title: A Study to Compare the Efficacy of an Extended-cycle Oral Contraceptive, Seasonique Which Utilizes Ethinyl Estradiol During the Usual Hormone-free Interval Compared to Conventional Oral Contraceptive Therapy for Cyclic Pelvic Pain
Brief Title: A Study to Evaluate the Efficacy of Seasonique for the Treatment of Cyclic Pelvic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Duramed Protocol Chair, Duramed Research, Inc.
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR-PSE-305
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Dysmenorrhea
Keywords: cyclic pelvic pain; dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Seasonique; Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: levonorgestrel/EE 0.15/0.03 and EE 0.01 mg tablets
- 2 (Active Comparator)
  Interventions: Drug: levonorgestrel/EE 0.15/0.03 mg tablets and placebo

INTERVENTIONS:
Drug: levonorgestrel/EE 0.15/0.03 and EE 0.01 mg tablets — 1 tablet daily
  Other Names: Seasonique
  Arms: 1
Drug: levonorgestrel/EE 0.15/0.03 mg tablets and placebo — 1 tablet daily
  Other Names: Portia
  Arms: 2

SUMMARY:
This study is being conducted to evaluate the effects of treatment with Seasonique an extended-regimen oral contraceptive that utilizes low dose ethinyl estradiol during the typical hormone-free interval. Patients will receive 26 weeks of treatment. The overall study duration will be approximately 9 months. Patients will be required to record menstrual pain in a daily diary.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe menstrual-related pain
* Regular spontaneous menstrual cycles

Exclusion Criteria:

* Any contraindication to the use of oral contraceptives
* Treatment with an oral contraceptive in the last 3 months
* Previous treatment failure with an extended oral contraceptive regimen

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2005-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the clinical assessment of dysmenorrhea | Baseline to Week 4,8,12,24, and 26 or early discontinuation

SECONDARY OUTCOMES:
Change from baseline in clinical assessment of dysmenorrhea (assessment of 4 additional symptoms) | Baseline to Weeks 4, 8, 12, 24 and 26 or early discontinuation
Incidence of menstrual bleeding and/or spotting | Duration of study
Analgesic use | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Protocol Chair, Study Chair — Duramed Research, Inc.
Locations (17):
- United States (17):
  - Duramed Investigational Site, Huntsville, Alabama
  - Duramed Investigational Site, Phoenix, Arizona
  - Duramed Investigational Site, San Diego, California
  - Duramed Investigational Site, Denver, Colorado
  - Duramed Investigational Site, Tampa, Florida
  - Duramed Investigational Site, Decatur, Georgia
  - Duramed Investigational Site, Moorestown, New Jersey
  - Duramed Investigational Site, Charlotte, North Carolina
  - Duramed Investigational Site, Columbus, Ohio
  - Duramed Investigational Site, Medford, Oregon
  - Duramed Investigational Site, Philadelphia, Pennsylvania
  - Duramed Investigational Site, Memphis, Tennessee
  - Duramed Investigational Site, Salt Lake City, Utah
  - Duramed Investigational Site, Newport News, Virginia
  - Duramed Investigational Site, Norfolk, Virginia
  - Duramed Investigational Site, Spokane, Washington
  - Duramed Investigational Site, Tacoma, Washington